CLINICAL TRIAL: NCT02402595
Title: A Phase 1, Single-center, Randomized, Double-blind, Double-dummy, Drug Interaction Study Between AVP-923 and Itraconazole, and Between AVP-786 and Itraconazole in Healthy Adult Subjects
Brief Title: Drug Interaction Study Between AVP-923 and Itraconazole and Between AVP-786 and Itraconazole in Healthy Adult Subejcts
Acronym: DDI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Avanir Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 15-AVP-786-103
Record Dates: First submitted 2015-02-26; First posted 2015-03-30 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Healthy
Keywords: Drug-drug interaction; Healthy Volunteers; Pharmacokinetics; deuterated dextromethorphan; dextromethorphan; dextromethorphan with quinidine; deuterated dextromethorphan with quinidine; itraconazole
MeSH Terms: interventions — dextromethorphan - quinidine combination; Itraconazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sequence 1 - Period 1 (Experimental): AVP-923 and placebo matching AVP-786- BID Day 1 until am of Day 15 Itraconazole - 200 mg BID on Day 9 followed by QD dosing on Days 10-15
  Interventions: Drug: AVP-923; Drug: Itraconazole
- Sequence 1 - Period 2 (after 3-week washout) (Experimental): AVP-786 and placebo matching AVP-923 - BID on Day 1 until am of Day 15 Itraconazole - 200 mg BID on Day 9 followed by QD dosing on Days 10-15
  Interventions: Drug: AVP-786; Drug: Itraconazole
- Sequence 2 - Period 1 (Experimental): AVP-786 and placebo matching AVP-923 - BID on Day 1 until am of Day 15 Itraconazole - 200 mg BID on Day 9 followed by QD dosing on Days 10-15
  Interventions: Drug: AVP-786; Drug: Itraconazole
- Sequence 2 - Period 2 (after 3-week washout) (Experimental): AVP-923 and placebo matching AVP-786- BID on Day 1 until am of Day 15 Itraconazole - 200 mg BID on Day 9 followed by QD dosing on Days 10-15
  Interventions: Drug: AVP-923; Drug: Itraconazole

INTERVENTIONS:
Drug: AVP-923
  Arms: Sequence 1 - Period 1; Sequence 2 - Period 2 (after 3-week washout)
Drug: AVP-786
  Arms: Sequence 1 - Period 2 (after 3-week washout); Sequence 2 - Period 1
Drug: Itraconazole
  Other Names: Sporanex

SUMMARY:
The purpose of this study is to determine the effects of a potent CYP3A4 inhibitor, itraconazole, on the steady-state PK of AVP-923 and AVP-786.

DETAILED DESCRIPTION:
A Phase 1, single-center, randomized, double-blind, double-dummy drug interaction study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males and females, 18 to 55 years of age
* Body Mass Index (BMI) ≥19 and ≤30 kg/m2 (for both males and females)

Exclusion Criteria:

* History or presence of significant disease
* History of substance abuse or dependence (except caffeine), or treatment for substance use disorder(s) within the year prior to screening or within 6 months for nicotine including e-cigarettes
* Use of any tobacco-containing or nicotine-containing products within 6 months prior to the first dose
* Use of any prescription or the over-the-counter medications within 14 days

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in plasma concentration of AVP-923 after dosing in combination with itraconazole | 16 Days
Change in plasma concentration of AVP-786 after dosing in combination with itraconazole | 16 Days

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) for AVP-923 and itraconazole | 16 Days
Incidence of adverse events (AEs) for AVP-786 and itraconazole | 16 Days

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kankam, MD, PhD, MPH, Principal Investigator — Vince and Associates Clinical Research Inc.
Locations (1):
- Vince and Associates Clinical Research, Inc., Overland Park, Kansas, United States